CLINICAL TRIAL: NCT01545323
Title: Phase I Study of Ex-vivo Lentiviral Gene Therapy for the Inherited Skin Disease Netherton Syndrome
Brief Title: Gene Therapy for Netherton Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10MI30
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Netherton Syndrome
Keywords: Netherton syndrome; Gene therapy; SPINK5
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One 20cm2/10cm2 autologous skin sheet graft (Experimental): Adults will receive a graft of approximately 20cm2. Children under 16 years of age will receive a graft around half this size, around 10cm2 .The graft is derived from SPINK5 transduced cells
  Interventions: Genetic: One 20cm2/10cm2 autologous skin sheet graft

INTERVENTIONS:
Genetic: One 20cm2/10cm2 autologous skin sheet graft — Adults will receive a graft of approximately 20cm2. Children under 16 years of age will receive a graft around half this size, around 10cm2 .The graft is derived from SPINK5 transduced cells

SUMMARY:
Netherton Syndrome is a serious skin disorder caused by damage in a gene called SPINK5. This gene controls the formation of a protein called LEKTI, which important for skin barrier function. LEKTI inhibits certain enzymes (serine proteinases) in the outermost layer of the skin (epidermis). The function of the serine proteinases is to break down the intracellular cement that holds together the horny cells in the epidermis, in order for the skin to be able to shed cells (known as cell desquamation). LEKTI deficiency leads to an uninhibited desquamation of horny cells, and as a result the skin becomes red and scaly. The barrier function of the skin is also affected. The permeability of the skin increases, and its capacity to bind water decreases, which causes dryness. The thinness of the barrier also results in over absorption of chemicals, for example topical medical treatments. Historically one in ten infants dies before their first birthday. Currently there are no proven treatments to cure this condition.

The investigators have been developing a gene therapy approach to treat this disorder. The investigators have used a disabled virus (vector) to carry a functional copy of the SPINK5 gene into skin stem cells. Proof-of-principle experiments have shown the investigators can restore almost normal shape and size of the upper layer of the skin in skin grafts grown in the lab. Even if only a small number of cells are genetically modified to carry the corrected SPINK5 gene, there seems to be a correction over a wide area of the graft.

In this trial the investigators propose grafting of autologous epidermal sheets generated from genetically modified skin stem cells for the treatment of patients with Netherton Syndrome. The investigators anticipate production and release of LEKTI protein from even a small patch of skin will be beneficial.

DETAILED DESCRIPTION:
Netherton Syndrome is a serious skin disorder caused by damage in a gene called SPINK5. This gene controls the formation of a protein called LEKTI, which important for skin barrier function. LEKTI inhibits certain enzymes (serine proteinases) in the outermost layer of the skin (epidermis). The function of the serine proteinases is to break down the intracellular cement that holds together the horny cells in the epidermis, in order for the skin to be able to shed cells (known as cell desquamation). LEKTI deficiency leads to an uninhibited desquamation of horny cells, and as a result the skin becomes red and scaly. The barrier function of the skin is also affected. The permeability of the skin increases, and its capacity to bind water decreases, which causes dryness. The thinness of the barrier also results in over absorption of chemicals, for example topical medical treatments. Historically one in ten infants dies before their first birthday. Currently there are no proven treatments to cure this condition.

The investigators have been developing a gene therapy approach to treat this disorder. The investigators have used a disabled virus (vector) to carry a functional copy of the SPINK5 gene into skin stem cells. Proof-of-principle experiments have shown the investigators can restore almost normal shape and size of the upper layer of the skin in skin grafts grown in the lab. Even if only a small number of cells are genetically modified to carry the corrected SPINK5 gene, there seems to be a correction over a wide area of the graft.

In this trial the investigators propose grafting of autologous epidermal sheets generated from genetically modified skin stem cells for the treatment of patients with Netherton Syndrome. The investigators anticipate production and release of LEKTI protein from even a small patch of skin will be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SPINK5 mutations in both alleles by direct DNA sequencing
* Absence of LEKTI protein expression in the skin by in situ immunostaining
* Patient informed consent, or parental/guardian consent in the case of minor participant

Exclusion Criteria:

* History of skin malignancy or evidence of current active malignant skin disease
* Pregnancy
* Hepatitis A, B, C or HIV positive
* Current antibiotic resistant bacterial colonisation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Safety of gene modified grafts | 1 year
  Adverse events will be monitored and assessed throughout the duration of the trial. Patients will be followed-up on-trial for 1 year. Subsequently, patients will be followed-up off-trial for life, as part of normal clinical care.
Histological evidence of correction of graft skin architecture | 1 year
  A skin biopsy will be taken from the graft area to determine correction of the skin architecture and to identify expression of LEKTI at time points 1, 3, 6 & 12 months post-grafting.

SECONDARY OUTCOMES:
Detection of increased LEKT1 staining at site outside the graft | 1 year
  A skin biopsy will be taken from the graft area to enable LEKTI staining at time points 1, 3, 6 & 12 months post-grafting.
Immune response to graft/transgene | 1 year
  ELISPOT will be used to detect possible cell mediated responses against the gene modified graft at time points 1, 3, 6 & 12 months post-grafting.

CONTACTS AND LOCATIONS:
Overall Officials: Jemima Mellerio, Dr, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Jemima Mellerio, Dr, Principal Investigator — Guy's and St thomas Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas NHS Trust, London
  - Great Ormond Street Hospital for Children NHS Trust, London

REFERENCES:
- [Background] Bitoun E, Micheloni A, Lamant L, Bonnart C, Tartaglia-Polcini A, Cobbold C, Al Saati T, Mariotti F, Mazereeuw-Hautier J, Boralevi F, Hohl D, Harper J, Bodemer C, D'Alessio M, Hovnanian A. LEKTI proteolytic processing in human primary keratinocytes, tissue distribution and defective expression in Netherton syndrome. Hum Mol Genet. 2003 Oct 1;12(19):2417-30. doi: 10.1093/hmg/ddg247. Epub 2003 Jul 29. PMID 12915442
- [Background] Chavanas S, Bodemer C, Rochat A, Hamel-Teillac D, Ali M, Irvine AD, Bonafe JL, Wilkinson J, Taieb A, Barrandon Y, Harper JI, de Prost Y, Hovnanian A. Mutations in SPINK5, encoding a serine protease inhibitor, cause Netherton syndrome. Nat Genet. 2000 Jun;25(2):141-2. doi: 10.1038/75977. PMID 10835624
- [Derived] Di WL, Mellerio JE, Bernadis C, Harper J, Abdul-Wahab A, Ghani S, Chan L, Martinez-Queipo M, Hara H, McNicol AM, Farzaneh F, McGrath J, Thrasher A, Qasim W. Phase I study protocol for ex vivo lentiviral gene therapy for the inherited skin disease, Netherton syndrome. Hum Gene Ther Clin Dev. 2013 Dec;24(4):182-90. doi: 10.1089/humc.2013.195. PMID 24329107